CLINICAL TRIAL: NCT03325673
Title: Randomized, Double-arm, Controlled Clinical Trial to Evaluate the Symptoms in Symptomatic Contact Lens Wearers Following Application of Intranasal Tear Neurostimulator Versus Control (CORIANDER)
Brief Title: Clinical Trial to Evaluate the Symptoms in Symptomatic Contact Lens Wearers Following Application of Intranasal Tear Neurostimulator Versus Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OCUN-024
Record Dates: First submitted 2017-10-03; First posted 2017-10-30 (Actual); Results first posted 2019-12-06 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TrueTear (Experimental): TrueTear Device (Intranasal Tear Neurostimulator) was used intranasally on contact lens (CL) wear days; it was also used on non-CL wear days if the participant chose. The number of applications was determined by participant.
  Interventions: Device: TrueTear
- TrueTear Sham Control (Sham Comparator): TrueTear sham device, which is not electrically active and has limited tip insertion depth, was used intranasally on CL wear days; it was also used on non-CL wear days if participant chose. The number of applications was determined by participant.
  Interventions: Device: TrueTear Sham Control

INTERVENTIONS:
Device: TrueTear — TrueTear Device (Intranasal Tear Neurostimulator) was used intranasally on CL wear days; it was also used on non-CL wear days if the participant chose. The number of applications was determined by participant.
  Arms: TrueTear
Device: TrueTear Sham Control — TrueTear sham device, which is not electrically active and has limited tip insertion depth, was used intranasally on CL wear days; it was also used on non-CL wear days if participant chose. The number of applications was determined by participant.
  Arms: TrueTear Sham Control

SUMMARY:
This study will evaluate the increase in comfort and comfortable contact lens (CL) wear time associated with application of TrueTear (active intranasal neurostimulation) compared with application of TrueTear sham control (intranasal application which is not electrically active) in symptomatic CL wearers.

ELIGIBILITY:
Inclusion Criteria:

A person is eligible for inclusion if he/she

* In at least one eye, has a cotton swab nasal stimulation Schirmer test score at least 4 mm greater than 3 minute Schirmer with anesthesia basal score in the same eye at the Screening Visit
* Is an adapted soft contact lens wearer and currently wears lenses an average of at least 2 days per week, with an average minimum wearing time of 3 hours each day over the past month and is able and willing to wear lenses for at least 6 hours on four study day visits
* Has at least 20/40 visual acuity in both eyes with CL correction
* Is symptomatic according to Young's categorization

Exclusion Criteria:

* Refractive error surgery
* Chronic or recurrent epistaxis, coagulation disorders or other conditions that may increase the risk of bleeding
* History of nasal or sinus surgery
* Vascularized polyp, deviated septum or severe nasal airway obstruction at the Screening visit
* Cardiac demand pacemaker, implanted defibrillator, or other active implanted metallic or active implanted electronic device in the head

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Senchyna, Study Chair — Allergan
Locations (1):
- Centre for Contact Lens Research School of Optometry & Vision Science, University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- TrueTear Sham Control: TrueTear sham device, which is not electrically active and has limited insertion depth, was used intranasally on CL wear days; it was also used on non-CL wear days if participant chose. The number of applications was determined by participant.
Period: Overall Study
Arm/Group | TrueTear | TrueTear Sham Control
Started | 42 | 42
Completed | 38 | 42
Not Completed | 4 | 0
Not completed — Adverse Event | 4 | 0

BASELINE CHARACTERISTICS:
Population: All eligible participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | TrueTear | TrueTear Sham Control | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (9) | 27 (9) | 28 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 32 | 67
  Male | 7 | 10 | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Contact Lens Dry Eye Questionnaire (CLDEQ-8) Score in the Study Eye
Description: The CLDEQ-8 is a validated questionnaire used to quantify symptoms experienced by the contact lenses (CLs) wearer. The participants were asked to respond to 8 questions about how their CLs performed over the preceding 2-week period. 4 questions (Eye discomfort, Eye dryness, Changeable blurry vision and Closing your eyes) answered on a scale of 0=Never to 4=Constantly; 3 questions about the end of wearing time (Discomfort, Dryness, Changeable blurry vision) answered on a scale of 0=Never have it to 5=Very Intense and 1 question (Removing your lenses) on a scale of 1=Never to 6=Several times a day for a total possible score of 1(best) to 37 (worst). The study eye was defined as the qualified eye with the greatest increase in tear production with stimulation by a cotton swab at the Screening Visit. If both eyes qualified, then the right eye was designated as the study eye.
Time Frame: Day 28
Population: All eligible participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TrueTear | TrueTear Sham Control
Number analyzed (Participants) | 38 | 40
score on a scale | 15.3 (5.6) | 17.2 (5.2)
Statistical Analysis 1: Comparison: TrueTear vs TrueTear Sham Control; Test type: Superiority; p = 0.116, Independent t-test

2. Primary Outcome: Comfort Rating Score in the Study Eye
Description: The participant assessed contact lens comfort in the study eye using a 100 point scale where a score of 0=Extremely uncomfortable and a score of 100=Extremely comfortable. The study eye was defined as the qualified eye with the greatest increase in tear production with stimulation by a cotton swab at the Screening Visit. If both eyes qualified, then the right eye was designated as the study eye.
Time Frame: CL Insertion, After 2 hours and the End of Day on Day 24
Population: All eligible participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TrueTear | TrueTear Sham Control
Number analyzed (Participants) | 38 | 40
score on a scale
  Insertion | 88 (11) | 86 (16)
  After 2 hours: number analyzed (Participants) | 37 | 39
  After 2 hours | 86 (11) | 82 (17)
  End of Day 24: number analyzed (Participants) | 35 | 36
  End of Day 24 | 75 (17) | 69 (19)
Statistical Analysis 1: Comparison: TrueTear vs TrueTear Sham Control; Insertion; Test type: Superiority; p = 0.468, t-test, 2 sided
Statistical Analysis 2: Comparison: TrueTear vs TrueTear Sham Control; After 2 hours; Test type: Superiority; p = 0.235, t-test, 2 sided
Statistical Analysis 3: Comparison: TrueTear vs TrueTear Sham Control; End of Day; Test type: Superiority; p = 0.152, t-test, 2 sided

3. Primary Outcome: Comfortable Wear Time (CWT) in the Study Eye
Description: CWT was calculated by taking the difference between the time participants reported started to find their CLs getting uncomfortable and the reported insertion time for that day. The study eye was defined as the qualified eye with the greatest increase in tear production with stimulation by a cotton swab at the Screening Visit. If both eyes qualified, then the right eye was designated as the study eye.
Time Frame: Day 24
Population: All eligible participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TrueTear | TrueTear Sham Control
Number analyzed (Participants) | 34 | 36
minutes | 618 (272) | 574 (254)
Statistical Analysis 1: Comparison: TrueTear vs TrueTear Sham Control; Test type: Superiority; p = 0.488, t-test, 2 sided

4. Primary Outcome: Total Wear Time (Total WT) in the Study Eye
Description: Total WT was calculated by taking the difference between the time participants reported removing their CLs and the reported insertion time for that day. The study eye was defined as the qualified eye with the greatest increase in tear production with stimulation by a cotton swab at the Screening Visit. If both eyes qualified, then the right eye was designated as the study eye.
Time Frame: Day 24
Population: All eligible participants with data available for analysis at the given time-point.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | TrueTear | TrueTear Sham Control
Number analyzed (Participants) | 34 | 36
minutes | 747 (201) | 652 (233)
Statistical Analysis 1: Comparison: TrueTear vs TrueTear Sham Control; Test type: Superiority; p = 0.072, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Day 0 to Day 28 +/- 3 days
Arm/Group | TrueTear | TrueTear Sham Control
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 3/42 | 4/42
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TrueTear (N=42) | TrueTear Sham Control (N=42)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Headache (Nervous system disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-26): https://cdn.clinicaltrials.gov/large-docs/73/NCT03325673/Prot_SAP_000.pdf